CLINICAL TRIAL: NCT00023023
Title: A Prospective Study of Transfusion-Transmitted Infections
Brief Title: Study of Transfusion-Transmitted Infections
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 010231; 01-CC-0231
Record Dates: First submitted 2001-08-18; First posted 2001-08-20 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-06-11

CONDITIONS: Viral Disease; Blood Donation; Transfusion-Transmitted Infections
Keywords: Hepatitis; Blood Bank; Viruses; Blood Donors; Blood Recipients; Natural History
MeSH Terms: conditions — Virus Diseases; Transfusion Reaction; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults and children subjects: The NIH and SH components will enroll and follow only adult (age >=18) blood donor or recipient subjects. CNMC will enroll and follow children between the ages of 6 months and 18 years.

SUMMARY:
This study will follow blood transfusion recipients for 6 to 9 months following transfusion to monitor the quality and safety of blood transfusion. Improved viral testing and careful donor screening in the last several years has dramatically reduced the rates of transfusion-related HIV and hepatitis. Nevertheless, ongoing surveillance of transfusion-related infections is essential to maintain a high safety standard and to determine the transfusion risk of other infectious agents, such as cytomegalovirus, Epstein-Barr virus, parvovirus B-19, HHV-8 (Kaposi s sarcoma virus) and other possible hepatitis viruses that might be blood-transmitted. Transfused patients blood will be tested for various infectious agents. Their blood samples and blood samples from their donors will be frozen and stored in a repository so that any new infectious agent can be rapidly evaluated for its danger to the safety of the blood supply.

Adult patients at the National Institutes of Health and children at the Children s National Medical Center who are scheduled to receive a blood transfusion or to undergo surgery for which a blood transfusion may be needed are eligible for this study.

All participants will have a 20- to 25-milliliter (about 2 tablespoonfuls) blood sample drawn before their transfusion and again at 1, 2, 4, 12 and 24 weeks after the transfusion. Patients who are transfused on more than one occasion over the course of the study will provide three additional monthly samples. Patients who develop a transfusion-transmitted infection during the study will provide up to four more samples to study the infection and its effects. Participants will complete a brief questionnaire at the end of the study regarding prior blood transfusions and the development of any illnesses, such as hepatitis, that might have been caused by the transfusion.

DETAILED DESCRIPTION:
Improved viral screening assays and more intensive questioning of donors for high-risk behaviors have resulted in dramatic declines in the rates of transfusion-transmitted hepatitis and AIDS. Nonetheless, there is need for continued vigilance of the safety of blood supply. This study will enroll blood donors and prospectively followed blood recipients in order to: 1) establish ongoing surveillance of the incidence of breakthrough infections from transfusion-transmitted agents for which there are existing donor-screening assays (e.g. HBV, HCV, HIV, human T cell lymphotropic virus [HTLV]); 2) monitor the transfusion risk of established infectious agents that are not routinely screened in blood donors including CMV, parvovirus B-19, and HHV-8 [Kaposi's sarcoma virus]; 3) establish a repository of linked donor and recipient samples so that any newly emerging infectious agent can be rapidly evaluated for its threat to the blood supply.

The risk of these blood transmitted infectious agents will be assessed by molecular and serologic assays in adult patients at NIH and Suburban Hospital in children at Children's National Medical Center. Blood samples from recipients transfused on one occasion will be obtained pre-transfusion and 1, 2, 4, 12, and 24 weeks post-transfusion. Recurrently transfused patients will have additional samples at 16 and 20 weeks after the index transfusion and 24 weeks after the last eligible transfusion. After initial infectious disease testing, recipient samples and linked donor samples will be stored in an off-site biorepository. The availability of the repository will allow for the assessment of transfusion risk for newly emerging pathogens and also for known agents for which there is no practical assay currently available. For example, this would allow future testing for prions in new variant Creutzfeld-Jacob disease (human variant of mad cow disease) or testing for the trypanosome that causes Chagas disease. Informed consent will be obtained to store and later test samples in the repository. Testing will be limited to infectious agents that potentially threaten the blood supply. No genetic testing will be performed.

ELIGIBILITY:
* INCLUSION CRITERIA

All adult (greater than or equal to 18 years) patients who are transfused at NIH will be eligible if:

1. they have not been transfused in the 6 weeks preceding the index transfusion;
2. they are expected to remain in the continental USA for at least six months post the index transfusion; and
3. if they are consented and a pre-sample is obtained
4. if they receive a transfusion during their NIH stay

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Under an established collaborative agreement and IRB authorization agreement between NIH and Suburban Hospital/Johns Hopkins Health System (JHHS), TRIPS will enroll patients undergoing open heart surgery at SH.
Sampling Method: Non-Probability Sample
Enrollment: 1771 (Actual)
Dates: Start 2002-01-17 (Actual)

PRIMARY OUTCOMES:
Positive viral DNA or RNA result | 1, 2, and 4 wk post-Txn
  Patients tests positive for any number of viral RNA/DNA which could infer transfusion-transmission.
Positive viral antibody result | 12, 24 and/or 6mo
  Patients tests positive for any number of viral antibodies which could infer transfusion-transmission.

SECONDARY OUTCOMES:
Viral discovery | 1, 2, and 4 wk and 12, 24 and/or 6mo
  Pre- and post- transfusion samples can be used for viral discovery programs employing GWAS, full genome sequencing or other methods that may evolve.

CONTACTS AND LOCATIONS:
Overall Officials: Valeria De Giorgi, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (3):
- United States (3):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - NIH Heart Center at Suburban Hospital Johns Hopkins Medicine, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- [Background] Schreiber GB, Busch MP, Kleinman SH, Korelitz JJ. The risk of transfusion-transmitted viral infections. The Retrovirus Epidemiology Donor Study. N Engl J Med. 1996 Jun 27;334(26):1685-90. doi: 10.1056/NEJM199606273342601. PMID 8637512
- [Background] Kleinman S, Busch MP, Korelitz JJ, Schreiber GB. The incidence/window period model and its use to assess the risk of transfusion-transmitted human immunodeficiency virus and hepatitis C virus infection. Transfus Med Rev. 1997 Jul;11(3):155-72. doi: 10.1053/tmrv.1997.0110155. No abstract available. PMID 9243769
- [Background] Alter HJ, Houghton M. Clinical Medical Research Award. Hepatitis C virus and eliminating post-transfusion hepatitis. Nat Med. 2000 Oct;6(10):1082-6. doi: 10.1038/80394. No abstract available. PMID 11017126
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-CC-0231.html